CLINICAL TRIAL: NCT06731166
Title: Effectiveness of Video Monitoring and Care Transition for Heart Failure Patients (EVIT-HF): Randomized Clinical Trial
Acronym: EVIT-HF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Uberlandia (Other)
Collaborators: Federal University of Rio Grande do Sul (Other); Universidade Federal do Triangulo Mineiro (Other)
Responsible Party: Principal Investigator, OMAR PEREIRA DE ALMEIDA NETO, Head, Federal University of Uberlandia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ethics committee 5.568.868
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Heart Failure With Reduced Ejection Fraction (HFrEF)
Keywords: Heart Failure; Nursing Care; Clinical Trial; Telenursing
MeSH Terms: conditions — Heart Failure | interventions — Self Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Videomonitoring Group (Experimental): Videomonitoring by cardiovascular nursing
  Interventions: Behavioral: self-care
- Voice call group (No Intervention): Voice call by cardiovascular nurses

INTERVENTIONS:
Behavioral: self-care — Videomonitoring provide by cardiovascular nurses
  Arms: Videomonitoring Group

SUMMARY:
The goal of this clinical trial is to measure the effectiveness of video monitoring associated with the transition of care for patients with heart failure.

The main questions it aims to answer is: Is video monitoring superior to monitoring via audio calls in patients with heart failure?

Researchers will compare monitoring by video to a monitoring by audio to see if drug videomonitoring works to improve selfcare in heart failure and other outocomes.

Participants will:

intervention group receive video calls guided by cardiologist nurses at 7, 30, 60, 180 and 365 days after hospital discharge.

the control group will receive audio calls for data collection, at the same time mentioned.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older;
* Admitted for decompensated HFrEF
* Ejection fraction less than 40% confirmed by echocardiogram performed in the last 3 months
* Who access to a mobile device with internet access

Exclusion Criteria:

* heart transplant waiting list;
* who had undergone coronary artery bypass in the last 3 months ;
* who were in palliative care;
* who had a life expectancy of less than 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Self-Care Behaviors Assessed by the European Self-Care Scale in Patients with Heart Failure | 365 days after discharge
  European Self-Care Scale The European self-care scale consists of 12 questions with a single domain related to self-care behavior. Responses to each item range from 1, "I completely agree", to 5, "I completely disagree", following a five-point Likert scale. The total score is obtained by summing all the responses, which can range from 12 to 60. Low values indicate better self-care. The items concern the various self-care behaviors of patients with heart failure, such as checking daily weight (item 1), rest (items 2 and 7), seeking help from the healthcare team (items 3, 4, 5 and 8), fluid restriction (item 6), diet (item 9), medication adherence (item 10), flu vaccination (item 11) and exercise (item 12)

SECONDARY OUTCOMES:
Rate of Cardiovascular Mortality within 365 Days Post-Discharge | 365 days after discharge
  Number of patients with heart failure who died during the trial

OTHER OUTCOMES:
Hospitalization Rates for Heart Failure within 365 Days Post-Discharge | 365 days after discharge
  Number of hospitalization of patients with heart failure during the trial
Heart Failure Knowledge Assessed by the HF Knowledge Questionnaire | 365 days after discharge
  HF Knowledge Questionnaire The HF knowledge questionnaire consists of 14 questions related to domains such as knowledge of the appropriate diet in HF, knowledge about the amount of fluids ingested and weight control, knowledge about pharmacological and nonpharmacological treatment of HF and general knowledge about the disease. The knowledge score is determined by the sum of the number of correct answers: for the correct question, the patient gains one point, and for each incorrect answer, the patient loses one point. In this way, the score ranges from 0 to 14
Adherence to Heart Failure Treatment Regimens asseded by "Adherence to HF treatment instrument" | 365 days after discharge
  Adherence to HF treatment Adherence to HF treatment will be assessed by an instrument with 10 questions related to the use of prescribed medications, daily weight checks, salt intake, water intake and attendance at scheduled appointments and exams. Each question has 3 to 4 alternatives; for questions with 4 alternatives, the score varied from 0 to 4 points, and for questions with 3 alternatives, the score varied from 0 to 3 points. Therefore, the general adherence score could vary from 0 to 26 points. A minimum score of 18 points will be considered a cutoff point for patients adhering to treatment, corresponding to 70% adherence
Quality of Life Assessed by the Minnesota Living with Heart Failure Questionnaire (MLHFQ) | 365 days after discharge
  Quality of life in HF patients The quality of life of patients with HF will be assessed by the Minnesota Living with Heart Failure Questionnaire (MLHFQ), a disease-specific questionnaire for patients with HF, comprising 21 items rated on six-point Likert scales representing different degrees of impact of HF on quality of life, from 0 (none) to 5 (very much). It provides a total score (range 0-105, from best to worst quality of life), as well as scores for two dimensions, physical (8 items, range 0-40) and emotional (5 items, range 0-25). The other eight items (a total of 21) are considered only for the calculation of the total score
Cardiorespiratory Fitness Assessed by the Veterans Specific Activity Questionnaire (VSAQ) | 365 days after discharge
  Cardiorespiratory fitness Cardiorespiratory fitness will be assessed by the Veterans Specific Activity Questionnaire (VSAQ), a brief questionnaire that consists of a list of activities presented in a progressive order according to metabolic equivalents (METs). Participants are instructed to determine which activities would cause fatigue, shortness of breath, chest discomfort, or necessity of stopping due to exhaustion if performed for a few minutes. The VSAQ was scored as a whole number (1 to 13 METs) directly from the subject's response. The VSAQ score will be adjusted by age and METs following a regression equation to predict aerobic fitness: METs = 4.7 + 0.97 × VSAQ - 0.06 × age

CONTACTS AND LOCATIONS:
Overall Officials: OMAR DE ALMEIDA NETO, PhD, Principal Investigator — Federal University of Uberlandia

IPD SHARING:
Plan to Share IPD: No
After careful consideration, we have decided not to share the individual patient data (IPD) from this study. This decision was made based on privacy concerns, participant confidentiality, and the specifics of the informed consent, which does not explicitly include authorization for sharing individual data.
  Furthermore, the study involves sensitive data that could compromise participants' privacy, even with anonymization and de-identification processes. Ensuring the safety and well-being of participants remains our top priority, and therefore, we have opted not to make individual data available on public platforms or repositories.
  The aggregated results and conclusions of the study will be shared through scientific publications, conferences, and other appropriate platforms to ensure that the findings benefit the scientific community and society at large.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-15): https://cdn.clinicaltrials.gov/large-docs/66/NCT06731166/Prot_SAP_000.pdf